CLINICAL TRIAL: NCT04783506
Title: Characterizing Inflammatory Profiles and Suicidal Behavior in Adolescents
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor, Founding Director of Center for Depression Research and Clinical Care, University of Texas Southwestern Medical Center
Other Study IDs: STU-2020-1297
Record Dates: First submitted 2021-02-25; First posted 2021-03-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Suicide and Depression
Keywords: suicide attempt; suicidal behavior; healthy control; adolescent; observational; depression; suicidal idation; suicide; anxiety; PTSD; substance abuse; healthy teen; depressed teen; children; teenage
MeSH Terms: conditions — Suicide; Depression; Suicide, Attempted; Anxiety Disorders; Stress Disorders, Post-Traumatic; Substance-Related Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will collect biospecimen samples of blood, plasma, serum, PBMCs, DNA. Blood draws will be collected from participants at baseline and at 3 follow-up visits.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Suicidal Behavior: Adolescents who have suicidal behavior, which for this study, is defined by a recent (within 3 months of enrollment) suicide attempt or suicidal ideation warranting urgent evaluation.
  Interventions: Other: Observational Study
- At Risk for Mood Disorders: Adolescents at risk for mood disorders, which for this study, is defined by either personal history of anxiety disorder or substance use disorder or a history of trauma, or a first degree relative with a history of a mood disorder or suicidal history.
  Interventions: Other: Observational Study
- Healthy Control: Healthy adolescents with no lifetime history of any psychiatric or substance use disorders or a history of trauma. Additionally, no first-degree family member with a history of a mood disorder or suicidal history.
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study — There is no intervention provided by this study. Observed for 12-month period using questionnaires and study visits.

SUMMARY:
Despite increasing suicide rates in adolescents, there remains a paucity of approaches to use to prevent re-attempts. Any hope for breaking the code to prevent youth suicide lies in understanding biological factors that play a role. Evidence suggests that inflammation and immune system dysfunction may be linked to suicide. The investigators will develop immune profiles for adolescents with suicidal behavior and those at risk in order to develop tools that can be implemented for prevention efforts.

This study involves blood draws, answering questions, and completing questionnaires - no treatment or intervention is provided as part of this study. Participants will be screened to see if they qualify for this study using questionnaires.

Participants will be teens (ages 12-18 years) with recent suicidal behavior, teens at-risk for developing depression, and healthy control teens. Participants complete all study-related tasks four times over a period of 12 months. Electronic surveys will be sent to participants to complete monthly. Both the adolescent and if applicable, their parent (or legally authorized representatives, LARs), will answer questions regarding depression, anxiety, and suicidal thoughts/behaviors.

DETAILED DESCRIPTION:
The purpose of this study is to map inflammatory dysfunction to suicidal behavior and establish a reliable immune signature of suicide risk that can 1) guide future research into fundamental pathophysiology and 2) identify targets for drug development and guide clinical screening and risk management.

Background: In previous research, the investigators have identified targets of clinical utility for both suicide-risk identification and novel therapeutic development. Specifically, a state of immune hyper-reactivity that predisposes to suicidal behavior can be corrected by use of immunomodulatory agents.

Blood tests screening for presence of autoantibodies may be implemented as diagnostic tests to predict future suicide risk. Monoclonal antibodies have gained recent attention for their use in CNS disorders (such as multiple sclerosis and migraine) and have been shown to be effective for some patients with depression.

However, the utility of anti-inflammatory treatments for depression has been limited by a lack of biomarkers to guide their use. Thus, presence of autoantibodies may identify a sub-group of adolescents and young adults with suicidality who are candidates for treatment with monoclonal antibodies.

The investigators specifically hypothesize that depressed youths with suicide behavior have immune hyper-reactivity, as reflected in dysfunctional cells mediating both innate and adaptive immune response.

Study Items: Since this is an observational study, investigators will explore a comprehensive panel of carefully selected participant specific parameters: socio-demographic (age, ethnicity, economic); symptom severity measures (depressive symptoms, mood, and feelings); clinical (medical history, anxious depression, early life trauma), biological (biomarkers in blood), behavioral (cognitive, emotional), with the goal to develop the most robust predictive models of treatment response and of depression outcomes. There is no medication or non-medication treatment or intervention provided by this study.

ELIGIBILITY:
Inclusion Criteria

Study participants must:

1. Be adolescents (aged 12-18 years);
2. Have the ability to speak, read, and understand English. The parent(s) or legal guardians of minors must also speak, read and understand English;
3. Be willing to provide consent/assent. Consent will be provided by parents/LAR/guardian for youth under age 18 or by young adult participant, aged 18. Youth, aged 8-17, must be willing to provide assent;
4. Have the ability to complete clinical evaluations and self-report measures;
5. Meet criteria for one of these three groups:

   1. Adolescent with suicidal behaviors, defined as having a recent (within 3 months) suicide attempt or suicidal ideation warranting urgent evaluation;
   2. Adolescents at risk for mood disorders, defined by either personal history of anxiety disorder or substance use disorder or a history of trauma, or a first degree relative with a history of a mood disorder or suicidal history;
   3. Healthy adolescents with no lifetime history of any psychiatric or substance use disorders or a history of trauma. Additionally, no first-degree family member with a history of a mood disorder or suicidal history..

Exclusion Criteria

Study participants must not:

1. Have current poorly controlled asthma, acute/chronic infection or other medical condition(s) that may affect immune marker levels;
2. Have a current medication (e.g., corticosteroids) that may affect immune marker levels of reactivity;
3. Have any condition for which, in the opinion of the investigator or designee, study participation would not be in their best interest (including but not limited to cognitive impairment, unstable general medical condition, intoxication, active psychosis) or that could prevent, limit, or confound the protocol-specified assessments;
4. Be unable to provide a stable home address and contact information

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents with suicidal behavior, at risk for mood disorder, and/or healthy controls will be recruited from several sources. Some examples include existing pathways (i.e., patient population, participants of ongoing/previous longitudinal studies) as well as an open invitation to the public for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Comprehensively characterize inflammatory tone and response | Baseline
  This will be accomplished by characterization of cells that mediate immune response. Numbers of these cells in blood and how they respond to immune stimulation will be compared between groups of adolescents with varying levels of suicidal behavior.

SECONDARY OUTCOMES:
Quantify levels of autoantibodies | Baseline
  This will be accomplished by measurement of antibodies against a broad panel of autoantigen. Levels of these autoantibodies will be compared between groups of adolescents with varying levels of suicidal behavior.

OTHER OUTCOMES:
Stability of immune signatures | Baseline, Month 3, Month 6 and Month 12
  This will be accomplished by comparing the stability of immune markers between groups of adolescents with varying levels of suicidal behavior.
Assess immune cell characterization | Baseline, Month 3, Month 6 and Month 12
  This will be accomplished by utilizing whole blood samples for flow cytometry to assess a broad range of immune cell characterization, encompassing granulocytes, monocytes, lymphocytes to help identify putative clinical targets that would identify increased risk of and treatment for suicidality.
Predict Clinical Health Risk Tracking Scale, Self-report (CHRT-SR) total | Baseline, Month 3, Month 6 and Month 12
  This will be accomplished by predicting levels of CHRT-SR using levels of immune markers concurrently or at previous visits.

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar H Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided